CLINICAL TRIAL: NCT03241576
Title: Provision of Small vs. Large Portion Sizes and Later Self-selected Food Intake: 3 Experimental Laboratory Studies in UK Participants
Brief Title: Provision of Small vs. Large Portion Sizes and Later Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Senior Lecturer, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 463882A
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small portion size provision (Experimental): Participants in this arm are served a small serving of a lunchtime food to eat (session 1).
  Interventions: Behavioral: Small portion size provision
- Large portion size provision (Active Comparator): Participants in this arm are served a large serving of a lunchtime food to eat (session 1).
  Interventions: Behavioral: Large portion size provision

INTERVENTIONS:
Behavioral: Small portion size provision — The intervention is the small meal size participants are provided with during a lunchtime session in the laboratory.
  Arms: Small portion size provision
Behavioral: Large portion size provision — The intervention is the large meal size participants are provided with during a lunchtime session in the laboratory.
  Arms: Large portion size provision

SUMMARY:
In 3 laboratory experiments the effect that receiving a small vs. large portion size of food has on later intake of that food was examined

DETAILED DESCRIPTION:
Historical increases in the size of commercially available food products have been linked to the emergence of a worldwide obesity crisis. Although the acute effect portion size has on food intake is well established, the effect that exposure to smaller portion sizes has on future portion size selection is yet to be examined.We tested whether reducing a food portion size may 'renormalize' perceptions of what constitutes a normal amount of food to eat and result in people selecting and consuming smaller portions of that food in future. Across three experiments participants were served a large or smaller portion of food. In experiments 1-2, twenty four hours later participants freely selected and consumed a portion of that food. In experiment 3, one week later participants reported on their preferred portion size of that food.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* History of food allergy, eating disorder or currently dieting to lose weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Later food intake (24 hour) | Measured 24 hours after random allocation (experiments 1 and 2)
  Amount of the lunchtime food later chosen and consumed
Later food intake (7 days) | Measured 7 days after allocation (experiment 3)
  Amount of the lunchtime food later chosen and consumed

IPD SHARING:
Plan to Share IPD: Yes
Open science framework
Time Frame: From Publication onwards
Access Criteria: Openly available to all
URL: https://osf.io/agk2d/

REFERENCES:
- [Derived] Robinson E, Kersbergen I. Portion size and later food intake: evidence on the "normalizing" effect of reducing food portion sizes. Am J Clin Nutr. 2018 Apr 1;107(4):640-646. doi: 10.1093/ajcn/nqy013. PMID 29635503